CLINICAL TRIAL: NCT01698593
Title: Bupivacaine Digital Blocks: How Long is the Pain Relief and Temperature Elevation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lalonde, Donald H., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RS#2009-1356
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Pain
Keywords: Bupivacaine; digital nerve block; epinephrine; duration of action; pain; touch; pressure; temperature
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- Ring Finger Nerve Block (Active Comparator)
  Interventions: Drug: Bupivacaine 0.5%; Drug: Bupivacaine 0.5% + Epinephrine (1:200,000)

INTERVENTIONS:
Drug: Bupivacaine 0.5%
Drug: Bupivacaine 0.5% + Epinephrine (1:200,000)

SUMMARY:
No one knows how long bupivacaine finger blocks last. Many use bupivacaine with and without epinephrine, but no one knows how the epinephrine affects the duration of the block. We also don't know how long the pain part of the block lasts, which is what counts.

The goal of the study is to determine the duration of action of bupivacaine digital nerve blocks (with and without epinephrine) on finger temperature and the sensory modalities of pain, touch, and pressure. 2 ml of bupivacaine 0.5% with and without epinephrine will be injected at the base of each ring finger on the palm surface. At the end of 1 hr, 6 hrs, 12 hrs, 14 hrs and each additional hour, patients will use an insulin lancet to measure pain, the Semmes Weinstein monofilament test to measure light touch and pressure and a body surface thermometer to measure finger temperature. The time for the finger to return to normal sensation and temperature will be measured.

DETAILED DESCRIPTION:
Lidocaine finger blocks have been shown to provide analgesia for nearly 5 hours without epinephrine and approximately 10 hours with epinephrine - essentially doubling its duration.1,2 The analgesic effect of epinephrine on the duration of bupivacaine finger blocks remains unknown.

Bupivacaine finger injection provides a much longer duration of action than lidocaine. Previous studies have shown the duration of action to be as long as 24.9 hours.1 In the senior author's experience, however, patients who get bupivacaine blocks start asking for pain medication as early as 7 hours after the block. Is it possible that the pain blocking effect of bupivacaine has a different duration than the touch and pressure effects? The answer to this question also remains unknown.

The third unknown question about bupivacaine digital blocks is their effect on fingertip temperature. It has been shown that lidocaine wrist blocks increase temperature in finger tips, and this has been postulated to be potentially helpful in frostbite to provide pain relief and hyperemia.3 Previous studies have shown bupivacaine to exhibit vasodilatory properties at clinical concentrations of injection.4-7 Does bupivacaine provide increased warmth to the finger tip? How long does it last?

The goals of this study are three fold: 1.) To determine what effect epinephrine has on the duration of bupivacaine finger block anesthesia. 2.) To assess the duration of action of bupivacaine with and without epinephrine on the digital sensory modalities of pain, touch and pressure, and 3.) To assess the finger tip temperature changes that result from bupivacaine digital blocks with and without epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteer

Exclusion Criteria:

* Under the age of majority
* Unable to give consent
* Pregnancy
* Diabetes
* Allergy to local anesthetic
* Prior finger surgery
* Preexisting digital vascular ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Time to return of pin-prick (pain) sensation | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Saint John Regional Hospital, Saint John, New Brunswick, Canada